CLINICAL TRIAL: NCT01855334
Title: A Randomized, Controlled Trial of L-arginine and Spironolactone in Dialysis-dependant End Stage Renal Disease
Brief Title: L-Arginine and Spironolactone Trial in Dialysis-Dependent ESRD
Acronym: LAST-D
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: change of funding leading to major redesign
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Joslin Diabetes Center (Other)
Responsible Party: Principal Investigator, David Charytan M.D., Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01DK096189
Record Dates: First submitted 2013-05-14; First posted 2013-05-16 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: End Stage Renal Disease; Hemodialysis
Keywords: Dialysis; ESRD; Cardiovascular disease; spironolactone; L-arginine; myocardial perfusion; coronary flow reserve; diastolic function
MeSH Terms: conditions — Kidney Failure, Chronic; Cardiovascular Diseases | interventions — Spironolactone; Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Spironolactone + Placebo (Experimental): Spironolactone 25 mg by mouth daily + Placebo L-arginine-liquid formulation by mouth 3 times daily
  Interventions: Drug: Spironolactone; Drug: Placebo
- Double Placebo (Placebo Comparator): Placebo spironolactone-1 tablet by mouth daily + Placebo L-arginine liquid formulation by mouth 3 times daily
  Interventions: Drug: Placebo
- Spironolactone + L-arginine (Experimental): Spironolactone 25 mg daily + L-arginine 3 grams orally 3 times daily
  Interventions: Drug: Spironolactone; Dietary Supplement: L-arginine
- L-arginine + Placebo (Experimental): L-arginine 3 grams by mouth 3 times daily + Placebo spironolactone 1 tablet by mouth daily
  Interventions: Dietary Supplement: L-arginine; Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone
  Other Names: Aldactone
  Arms: Spironolactone + L-arginine; Spironolactone + Placebo
Dietary Supplement: L-arginine
  Arms: L-arginine + Placebo; Spironolactone + L-arginine
Drug: Placebo
  Arms: Double Placebo; L-arginine + Placebo; Spironolactone + Placebo

SUMMARY:
Cardiovascular disease is the primary cause of death in patients with end stage renal disease (ESRD). New research suggests that the high risk of death may be partly due to high levels of fibrosis and a loss of small blood vessels in the heart of patients with dialysis-dependent ESRD. This study is designed to compare the effects of two different drugs, spironolactone and L-arginine, with placebo on structure and function of the heart in individuals with dialysis-dependent ESRD.

DETAILED DESCRIPTION:
We hypothesize that that abnormalities in aldosterone and nitric oxide (NO) homeostasis contribute to the progression of microvascular disease and myocardial fibrosis in ESRD and that agents designed to restore normal aldosterone and NO homeostasis will improve microvascular and diastolic cardiac function in the heart of individuals with dialysis dependent ESRD. We will test 2 specific agents: The mineralocorticoid receptor blocker spironolactone; and L-arginine, an agent which improves NO bioavailability. Two specific aims will be addressed using a prospective, double-blinded, 2x2 factorial trial in dialysis dependent patients with ESRD. Subjects will be randomized to placebo, spironolactone plus placebo, L-arginine plus placebo, or combination spironolactone and L-arginine therapy. Diastolic cardiac function will be assessed using tissue Doppler index (TDI) determined mitral annular velocities (E') on LV echocardiography, and microvascular supply will be assessed using CFR-the ratio of hyperemic to resting myocardial blood flow-measured by positron emission tomography (PET) scans at baseline, 2 weeks and after 9 months of randomized therapy.

This randomized trial of spironolactone and L-arginine will provide important data about the contributions of aldosterone and NO to the pathogenesis of cardiovascular disease in ESRD, will demonstrate the therapeutic potential of L-arginine and spironolactone as as targeted cardiovascular therapies for use in ESRD, and will provide important insights into the underlying pathophysiology of cardiovascular disease in ESRD. The results generated will provide the data needed to design large-scale trials testing whether spironolactone or L-arginine can improve mortality or cardiovascular outcomes in ESRD.

ELIGIBILITY:
Inclusion Criteria:

* Chronic dialysis therapy for End Stage Renal Disease
* Age 21-85

Exclusion Criteria:

* Hyperkalemia requiring unscheduled dialysis within 3 months
* Pre-dialysis potassium ≥6.5 meq/L within 3 months
* Hypotension defined as SBP <100
* Recurrent intra-dialytic hypotension defined as recurrent cramping, light-headedness, or hypotension requiring infusion of saline or other intervention or otherwise limiting ability to achieve dry weight. Or SBP <80
* History of myocardial infarction
* History of coronary artery bypass surgery
* Non revascularized coronary disease >90%
* Mitral valve repair or replacement
* Severe mitral valve disease
* Renal transplant expected within 9 months
* Expected survival < 9 months
* Pregnant
* Prisoners
* Unable to provide consent
* Allergy to spironolactone or L-arginine
* Digitalis use
* 1st or 2nd degree heart block

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Change in coronary Flow Reserve (PET) | Between baseline and 9 months
  Coronary flow reserve will be measured using rest and stress 13N ammonia myocardial positron emission tomography (PET) at baseline and 9 months
Change in left ventricular diastolic function | Between baseline and 9 months
  Left ventricular diastolic function will be measured using mitral annular E' on tissue doppler index echocardiography at baseline and 9 months

SECONDARY OUTCOMES:
Association between coronary flow reserve (CFR) and tissue doppler index (E') | Baseline
Change in resting myocardial blood flow | Between baseline and 9 months
Change in left ventricular mass index | Between baseline and 9 months
Change in coronary vascular resistance | Between 0 and 9 months
Association between change in coronary flow reserve (CFR) and change in diastolic function-tissue doppler index (E') | Between baseline and 9 months
Change in early diastolic function (E') | Between baseline and 2 weeks
Combined cardiovascular safety | Up to 9 months
  Combined rate of death, myocardial infarction, stroke, or hospitalization
Cardiovascular death | Up to 9 months
Hyperkalemia | Up to 9 months
  Hyperkalemia requiring extra dialysis, adjustment in dialysate potassium, or discontinuation of therapy
Hypotension | Up to 9 months
  Symptomatic or intradialytic hypotension up to 9 months
Change in early coronary flow reserve | Between baseline and 2 weeks
Change in hyperemic myocardial blood flow | Between baseline and 9 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

REFERENCES:
- [Derived] Hasegawa T, Nishiwaki H, Ota E, Levack WM, Noma H. Aldosterone antagonists for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2021 Feb 15;2(2):CD013109. doi: 10.1002/14651858.CD013109.pub2. PMID 33586138